CLINICAL TRIAL: NCT03020342
Title: A New Biomarker for Detection of Minimal Residual Tumor in Hepatitis-B Virus Related Hepatocellular Carcinoma After Curative Therapies: The Cell-free Circulating HBV-host Chimera DNA Fragment
Brief Title: HBV-host cfDNA as Minimal Residual Tumor Marker for HBV-related HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201510056RINA
Record Dates: First submitted 2016-06-22; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; chimera DNA; circulating DNA; biomarker
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor (T) and non-Tumor (NT) tissue, and peripheral blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
Early stage HCC is treated by curative surgical resection or by local ablation (such as radio-frequency) as the current standard of care. The complete removal of clinical visible HCC is then confirmed by imaging by MRI or CT, or by a decline of tumor marker (AFP or PIVKA). However, despite an apparent complete removal of the HCC, those post-curative patients frequently develop tumor recurrence at a rate ranging 10-50% within the first year. The high rate of early HCC recurrence indicated a minimal residual HCC after the curative therapies in a significant proportion of patients. A better and more specific biomarker for detecting the residual HCC will improve the patients' prognosis prediction and therapeutic plan.

To detect the minimal residual HCC, a biomarker unique to the tumor is needed. Currently, the cell-free circulating DNA carrying tumor-specific somatic mutations has been advocated as a promising one. It has been applied to investigate the tumor responses or resistances to cancer therapy. However, currently it is restricted to detect or follow only large advanced cancer, because of the difficulty in separating or enriching the cfDNA with tumor-specific mutations from the cfDNA from normal cells. In this project, the investigators proposed that one class of somatic mutation in HBV-related HCC, namely the insertion mutagenesis by integrated HBV DNA, could be adopted to circumvent this difficulty. HBV DNA integration has been found in the chromosomes of about 90% of HBV-related HCC and the integration site is unique to individual HCC. The HBV-host junction DNA fragment from one HCC is therefore a tumor-specific biomarker. Such fragments can be released into the circulation as cell-free circulating DNAs, and the detection of the HBV-host chimera DNAs in the circulation is a reliable evidence for the presence of the tumor in the patient. Therefore the cf circulating HBV-host chimera DNA is proposed to assay any minimal residual HCC after curative therapies.

DETAILED DESCRIPTION:
Development stages:

Stage I: Identification of integrated HBV DNA sites in HBV-related HCC tissues. the investigators will develop either HBV-specific inverse PCRs or capture-sequencing protocols to identify HBV integrations sites in the tumor chromosomes. The viral-host junction sequences of individual HCC identified and used as the template for developing assays for detecting the same HBV-host chimera DNA fragment in the circulation.

Stage II: New platforms to accurately detect or even quantitate the circulating vh-chimera DNA fragment.

These tumor-specific vh-chimera DNA will only represent a tiny fraction of total cfDNAs. However, as these sequences of the tumor-specific vh-chimera DNA have been known from stage 1, the investigators may develop better and more specific assays for quantitation.

Stage III: Assays for cell-free tumor specific vh-chimera DNA applied to the blood samples from post-curative HCC patients.

To demonstrate the efficacy of these assays, blood samples obtained at 4 weeks after curative therapies from 50 HBV-related HCC patients, and tested for the presence of cf tumor-specific vh-chimera DNAs. The presence or absence of such vh-chimera DNA will be correlated with the early HCC recurrence within the first year to determine any clinical significance. There will be one blood sampling at the time of HCC recurrence.

Sample collection In stage I and II, the investigators will set up methods for chimera DNA identification and quantification, which need tumor samples to support the development and evaluation of the feasibility for each assay. Therefore, the investigators will apply the approval for use the tissues from the Taiwan Liver Cancer Network (TLCN), including 20 pairs of HBV-related male HCC, 20 pairs of HBV-related female HCC (for positive control), 20 pairs of HCV related male HCC, 20 pairs of HCV related female HCC (for negative control), 20 pairs of HBV- and HCV-related male HCC, and 20 pairs of HBV- and HCV-related female HCC (to see if vh-chimera DNA is also applicable for HBV- and HCV-related HCC). Both the genomic DNA and RNA will be applied for these 120 patients in total. Genomic DNA will be used in assay development, including identification, detection and quantification; whereas RNA will be used in validation of the insertional mutagenic RNA transcripts, which will provide supporting evidence for tumor specific integration from transcription level.

In stage III, the investigators will investigate whether there is any correlation between tumor-specific vh-chimera DNA level and recurrence-free survival using the assays the investigators developed in stage I and II. Therefore, the investigators will collect the Tumor (T) and non-Tumor (NT) tissue pairs from 50 HBV-related HCC patients that receive surgical removal of tumor, and also the peripheral blood at 4w after surgery. T and NT tissues are for vh-chimera DNA identification, peripheral blood will be used for vh-chimera DNA detection and quantification. On the other hand, clinical information including tumor size, tumor grade, serum markers from routine liver function test (ALT, AST), current HCC marker (AFP), and recurrence-free survival time will be collected for correlation study. All data will be stored in computer with password protection.

ELIGIBILITY:
Inclusion Criteria:

* HBV-related HCC patients that receive surgical removal of tumor.

Exclusion Criteria:

* unsuitable for surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV-related HCC patients that receive surgical removal of tumor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
vh-chimera DNA | week 4 after surgery.
  Detection of the HBV-host chimera DNA in blood sample.----- one blood sampling at the time of HCC recurrence.

SECONDARY OUTCOMES:
Tumor size (measured in the longest dimension in cm) | after medical imaging or pathology report completion, up to 2 weeks.
  clinical information about HCC recurrence. detection by CT or MRI.
tumor grade (Grades I-IV) | after medical imaging or pathology report completion, up to 2 weeks.
  clinical information about HCC recurrence. detection by CT or MRI.
recurrence-free survival time ----measurement in weeks | from the date of surgery until the date of first documented HCC recurrence or date of death from any cause, whichever came first, assessed up to 24 months
  clinical information about HCC recurrence.

OTHER OUTCOMES:
Routine liver function test (ALT in IU/L) | week 4 after surgery, ---- one blood sampling at the time of HCC recurrence.
  serum markers.
Routine liver function test (AST in IU/L) | week 4 after surgery, ---- one blood sampling at the time of HCC recurrence.
  serum markers.
current HCC marker (AFP ng/ml) | week 4 after surgery, ---- one blood sampling at the time of HCC recurrence.
  serum markers.(ALT and AFP)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, MD-PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided